CLINICAL TRIAL: NCT00809562
Title: An Exploratory Fixed Dose Randomized Double Blind Parallel-group Placebo-controlled Study of the Safety and of the Therapeutic Effects of Ro 4917523 in Patients With Treatment- Resistant Depression
Brief Title: A Study of RO4917523 in Patients With Treatment Resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP22022
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — 2-chloro-4-(1-(4-fluorophenyl)-2,5-dimethyl-1H-imidazol-4-ylethynyl)pyridine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: RO4917523
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — po daily for 10 days
  Arms: 2
Drug: RO4917523 — orally daily for 10 days, cohorts receiving up to 5 different doses (according to safety and tolerability)
  Arms: 1

SUMMARY:
This study will evaluate the safety, tolerability and efficacy of RO4917523, in comparison to placebo, in patients with treatment-resistant depression. Following a washout period from existing anti-depressant medication, cohorts of patients will be randomized to receive daily oral RO4917523 at up to five different doses (according to the safety and tolerability observed at the lower doses during the study), or placebo. The anticipated time on study treatment is 10 days (in an inpatient unit), and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-65 years of age;
* recurrent major depressive disorder, without psychotic features;
* at least 3 lifetime treatment failures, at least 2 of which must have occurred within the current depressive episode;
* baseline minimal severity defined by a HAM-D score of 18 or above;
* willing to be hospitalized for at least 16 consecutive days.

Exclusion Criteria:

* history of bipolar disorder, schizoaffective disorder or schizophrenia;
* history of psychosis, including psychotic depression;
* significant past or present neurological disorder, including seizures, stroke and/or head trauma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Adverse events, ECGs, laboratory parameters,vital signs | Throughout study

SECONDARY OUTCOMES:
Efficacy: MADRS score | From baseline to day 10
Symptoms of treatment-resistant depression | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- United States (7):
  - Oceanside, California
  - San Diego, California
  - New Haven, Connecticut
  - Shreveport, Louisiana
  - Flowood, Mississippi
  - New York, New York
  - Pittsburgh, Pennsylvania